CLINICAL TRIAL: NCT03266718
Title: A Couple-Based Physical Activity Intervention for Cancer Survivors
Brief Title: Move 2 Health: A Couple-Based Physical Activity Intervention for Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00060926
Record Dates: First submitted 2017-08-15; First posted 2017-08-30 (Actual); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Physical Activity; Cancer Survivor
Keywords: cancer survivor; breast cancer; prostate cancer; couples
MeSH Terms: conditions — Motor Activity; Breast Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Activity Intervention (Other): Couples will receive four 60-minute intervention sessions via videoconference with Duke staff. Study staff will provide couples with instructions for use of the iPad computer and videoconference software which will be used to deliver the intervention sessions.The first 3 sessions will be conducted weekly, with a booster session occurring approximately one month later.
  Interventions: Behavioral: Physical Activity Intervention
- Waitlist control (Other): Couples will have the option to receive the intervention after they complete the follow-up survey. This version of the intervention will not include the booster session, so will last approximately 1 month in total. If they choose to receive the intervention, they will be provided with a tablet computer if they do not have one.
  Interventions: Behavioral: Physical Activity Intervention

INTERVENTIONS:
Behavioral: Physical Activity Intervention — To develop and test a couple-based physical activity intervention among cancer survivors and their partners

SUMMARY:
This pilot study will develop and test a couple-based physical activity intervention among cancer survivors and their partners.

Aim 1: To determine the feasibility and acceptability of a couple-based physical activity intervention for cancer survivors. Feasibility will be quantified using rates of study eligibility, overall accrual, attrition, and adherence to the study protocol. Acceptability will be assessed via couples' ratings on a standardized measure of treatment effectiveness/ satisfaction, supplemented open-ended questions

Aim 2: To provide preliminary data on the effects of a couple-based physical activity intervention relative to a wait list control group on survivor outcomes (i.e., level of physical activity, quality of life, self-efficacy for achieving and maintaining physical activity goals, perceived partner support for physical activity, and quality of the survivor-partner relationship). The investigators hypothesize that the intervention will produce benefits in each of these domains.

Aim 3: To provide preliminary data on the effects of a couple-based physical activity intervention relative to a wait list control group on partner outcomes (i.e., partner's level of physical activity, self-efficacy for helping the survivor achieve and maintain physical activity goals, and quality of the survivor-partner relationship). The investigators hypothesize that the couple-based intervention will produce benefits in each of these domains.

DETAILED DESCRIPTION:
Background and Significance:

Physical activity (PA) is an essential part of cancer survivors' treatment plan as it helps prevent recurrence and improves cardiovascular fitness and downstream cardiovascular risk, the cause for most deaths in cancer survivors. Additional benefits of increasing PA include improvements in body composition, physical function, psychological outcomes, and quality of life. However, most survivors are not sufficiently active and would benefit from an intervention to promote PA. Prior PA interventions for cancer survivors have had mixed success. A recent systematic review identified 14 RCTs testing exercise interventions among sedentary cancer survivors and concluded that there was insufficient evidence that existing interventions are successful in achieving recommended levels of PA. In particular, there has been a lack of attention to psychosocial aspects of changing behavior, and to strategies that promote independent exercise behavior that can be maintained over time. Thus, it is clear that novel approaches to PA interventions are needed.

Design:

This is a two-arm randomized controlled trial to evaluate a couple-based physical activity (PA) intervention that systematically trains partners in skills to support the survivor in PA initiation and maintenance strategies.

Couples randomized to Arm 1 (the Couples-Based Physical Activity Intervention) will receive four 60-minute intervention sessions via videoconference with Duke staff. Study staff will provide couples with instructions for use of the iPad computer (if provided by the study) and videoconference software which will be used to deliver the intervention sessions. Couples will also be provided with contact information for technical support. The first 3 sessions will be conducted weekly, with a booster session occurring approximately one month later. The intervention will include components to (a) encourage couples' favorable outcome expectations about the benefits of working together to initiate and maintain increases in PA, (b) build their confidence that they can work together to accomplish their goals, and (c) help them identify and use communal strategies, such as couple communication and joint decision making about goals and plans for increasing physical activity, and working through barriers to making these changes. Finally, the intervention will incorporate important behavior change techniques that have been found to help people change their exercise behavior, such as goal setting, self-monitoring of behavior, and prompts for practice, adapting them to a communal coping approach. Treatment sessions will be audio recorded for QA purposes.

Those randomized to Arm 2 (waitlist control) will have the option to receive the intervention after they complete the follow-up survey. This version of the intervention will not include the booster session, so will last approximately 1 month in total. If they choose to receive the intervention, they will be provided with a tablet computer if they do not have one.

ELIGIBILITY:
Inclusion Criteria:

* Survivor participants are those who have been diagnosed with breast or prostate cancer, who are married or in a committed relationship and live with their partner, and who are sedentary (e.g., not undertaking dedicated physical activity on 3 or more days per week). Both survivors and their partners must be at least 18 years of age, be fluent in English, and be eligible and willing to participate.

Exclusion Criteria:

* We will exclude patients and/or partners with known metastatic disease, who are hearing impaired, who are deemed too sick to participate, who have a medical condition that prohibits them from prolonged walking, who are participating in another research study that promotes increased exercise, or who have evidence of unstable cognitive or mental health problems who cannot properly provide consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2016-09-26 (Actual); Study Completion 2016-12-11 (Actual)

PRIMARY OUTCOMES:
Feasibility of a couple-based physical activity intervention for cancer survivors as measured by a composite score of total number of couples screened and rates for non-eligibility. | 2 months after baseline survey
Feasibility of a couple-based physical activity intervention for cancer survivors as measured by a composite score of total number of couples screened and rates of refusal. | 2 months after baseline survey
Acceptability of a couple-based physical activity intervention for cancer survivors as measured by a composite score of total number of couples screened and rates for non-eligibility. | 2 months after baseline survey
Acceptability of a couple-based physical activity intervention for cancer survivors as measured by a composite score of total number of couples screened and rates of refusal. | 2 months after baseline survey

SECONDARY OUTCOMES:
Efficacy as measured by steps taken | 2 months after baseline survey
Quality of life as measured by surveys | 2 months after baseline survey
Self -efficacy for achieving and maintaining physical activity goals as measured by surveys | 2 months after baseline survey
Perceived partner support for physical activity as measured by surveys | 2 months after baseline survey
Quality of the survivor-partner relationship as measured by surveys | 2 months after baseline survey

CONTACTS AND LOCATIONS:
Overall Officials: Laura Porter, PhD, Principal Investigator — Duke University

IPD SHARING:
Plan to Share IPD: No
We will not share IPD unless requested by Duke Researchers only.